CLINICAL TRIAL: NCT06927037
Title: Immersive Physical Therapy in the NICU: Comparing Delivery Models to Improve Infant and Parent Outcomes
Brief Title: Immersive Physical Therapy in the Neonatal Intensive Care Unit (NICU)
Status: Not yet recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation for Physical Therapy Research (Other)
Responsible Party: Sponsor
Other Study IDs: 24-2424
Record Dates: First submitted 2025-04-03; First posted 2025-04-15 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Physical Therapy; NICU Infants
Keywords: Physical Therapy; NICU infants; Parental Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Usual Care: A retrospective group of infants whose data represent usual care
- Small Baby Unit: A group comprised of infants and their parents that represent implementation of a Small Baby Unit (SBU)
- Immersive Physical Therapy: A group comprised of infants and their parents that represent the small baby unit where parents are also asked to administer physical therapy techniques with their infants

SUMMARY:
To learn if and how the physical and occupational therapy program in the Newborn Critical Care Center helps parents with their stress levels and ability to meet the needs of their preterm infants.

DETAILED DESCRIPTION:
Composed of one retrospective group and two prospective groups. Each group will be defined based on the stage of enrollment, which will coincide with the rollout of two different standard-of-care initiatives in the hospital. These initiatives are determined outside of the study protocol. The retrospective group will be composed of infants that are under the current initiative. The small baby unit will then be implemented within the hospital site, and infants and parents enrolled at that time will reflect the impact of the small baby unit. The small baby unit will then transition into an immersive physical therapy model, and any infants and parents enrolled at that time will reflect the impact of this second-tier initiative.

ELIGIBILITY:
Infant Inclusion Criteria:

* <28 weeks gestation at birth
* born or transferred to UNC's Newborn Critical Care Center within the first 48 hours of life
* If in the SBU or Immersive PT groups: Must be cared for at certain UNC Hospital locations through at least 34 weeks postmenopausal age

Infant Exclusion Criteria:

* Has a high likelihood of transferring to an outside hospital
* Has a genetic abnormality, congenital neurological or musculoskeletal disorder

Maternal Inclusion Criteria:

* Is the biological parent
* Sex is female
* Understands English or Spanish Language
* Is at least 18 years of age

Maternal Exclusion Criteria:

* Is not the biological parent
* Sex is male
* Does not understand English or Spanish language
* Is under 18 years of age

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants and parents identified as part of the NICU at certain University of North Carolina (UNC) Hospital locations
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of physical therapy visits | From birth to hospital discharge, assessed up to 4 months of life
  The number of physical therapy visits to the infant's bedside per week, as noted in the medical record
Number of physical therapy minutes billed | From birth to hospital discharge, assessed up to 4 months of life
  The number of physical therapy minutes billed per week as noted in the medical record
Number of physical therapy interactions by parent | From birth to hospital discharge, assessed up to 4 months of life
  The number of times per week that mothers report doing physical therapy with their infant, with higher numbers indicating a greater dosage
Infant Motor Skills | Assessed at 34 to 36 weeks postmenstrual age
  Motor skills will be measured via the Test of Infant Motor Performance, a 42-item test of functional motor skills with age standards from 34 weeks post-menstrual age through 17 weeks post-term. Scores range from 0 to 142 with higher scores indicating better performance. Scores are transformed into an age standard based on performance.

SECONDARY OUTCOMES:
Degree of Parent-Therapist Contact | From birth to hospital discharge, assessed up to 4 months of life
  The number of times per week that the parent received education on physical therapy techniques as documented in clinical notes
Infant Neurobehavior | Assessed at 34 to 36 weeks postmenstrual age
  Neurobehavior will be measured via the NeoNatal Neurobehavioral Scales-II, a valid and reliable neurobehavioral assessment for high-risk infants across 13 different scales, including habituation, attention, arousal, self-regulation, and more. Due to the varied performance across these scales and their different ranges, it can be challenging to determine an overall exam response for each infant. Therefore, grouping response patterns into discrete profiles through latent profile analysis offers a simpler way to compare NNNS performance among infants.
Change in Maternal Stress | From birth to hospital discharge, assessed up to 4 months of life
  Maternal Stress will be measured via the Parent Stress Scale: NICU, a 26-item tool to assess parent stress in NICU that covers topics such as: Infant Appearance, Parental Role Alteration, Sights & Sounds. Scores range from 0 to 130 with higher scores indicating greater stress
Change in Parent Competence | From birth to hospital discharge, assessed up to 4 months of life
  Parent Competence will be measured via the Parent Sense of Competence Scale,17-item scale to assess change in the parent's sense of competence in infant care. Scores range from 17 to 102 with higher scores indicating higher sense of competence

CONTACTS AND LOCATIONS:
Overall Officials: Dana McCarty, PT, DPT, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No